CLINICAL TRIAL: NCT04419740
Title: What is the Impact of an E-tool Based Mindfulness Intervention on Psychological Outcomes Compared to no Intervention in Infertile Women Undergoing Assisted Reproductive Technique Treatments: A Randomized Controlled Study?
Brief Title: Impact of a Mindfulness Intervention on Infertile Women Undergoing Assisted Reproductive Technique Treatments
Acronym: EMOT-IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Isabelle Streuli, Principal investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMOT-IVF
Record Dates: First submitted 2019-12-11; First posted 2020-06-05 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based psychological intervention (Experimental): Patients allocated to the intervention group will receive an email with a link to a video and a pdf document. The video and the pdf document will introduce them to the principles and the practice of mindfulness. They will also receive an access code to an e-tool valid for 1 month. On this e-tool the patient will have access to short guided meditations both general and specific to infertility. They will be instructed to follow the "découverte" (discovery) program of 8 meditations of 10 minutes and then the program "désir de parentalité (wish to become a parent) of 13 minutes 15 meditations of 13 minutes each. Patients will be given access to all other meditations programs of PetitBambou and instructed to meditate with the program for at least 10-15 minutes on a daily basis.
  Interventions: Behavioral: Mindfulness based psychological intervention
- Standard care (No Intervention): The control group will have no additional intervention and will receive standard care in the institution. Women in all 3 study sites have access to counselling/psychological support with a trained professional before treatment initiation. During that consultation coping and stress reduction strategies are discussed.

INTERVENTIONS:
Behavioral: Mindfulness based psychological intervention — Women in the intervention group will have to use an application during 1 month. They will do meditation during 15 minutes each day.
  Arms: Mindfulness based psychological intervention

SUMMARY:
Infertility and its treatments can have a significant impact on women's psychological health. Anxiety has a negative impact on quality of life during treatment and can lead to withdrawal of care. the investigators would like to test the effectiveness of an application available via the Internet that offers daily exercises such as mindfulness meditation. Women in the "treatment" group will be instructed to practice meditation exercises using the 15-minute daily application during in vitro fertilization treatment until pregnancy testing. Women in the control group will have the standard care of the centre. The investigators will measure the effectiveness of the intervention on anxiety, depression, quality of life and mindfulness aspects. The investigators will also assess the impact on the chances of pregnancy and stress.

DETAILED DESCRIPTION:
Infertility is an unexpected and stressful life with emotional, social and sexual repercussions. Women undergoing assisted reproductive techniques (ART) exhibit high anxiety and/or depression scores during the pre-treatment period, during the course of treatment and during the 2 weeks waiting-time for the pregnancy test.

The impact of psychological distress on ART outcomes is debated. Several studies report a negative impact of stress on pregnancy rates after IVF whereas two meta-analyses report inconclusive results regarding the association between emotional distress and pregnancy outcomes after ART.

The success rates of ART, which are highly dependent on the woman's age, are low in women in their late reproductive years with the need of several ART treatments to achieve pregnancy. Moreover, ART is often the last resort treatment in couples that have undergone infertility investigations and other first-line treatments such as surgery, ovulation induction and/or stimulation with intra-uterine insemination. Couple need resilience in order to undergo repeated treatments. Psychological distress therefore has an impact on cumulative pregnancy rates over several ART treatments because of premature treatment discontinuation. Depressive symptoms at baseline have been shown to predict treatment "dropout" after only one cycle.

Preliminary evidence suggests that mind-body interventions, including mindfulness-based interventions and yoga, may be effective in reducing mental health difficulties such as anxiety and depression in infertile women undergoing treatments.

The aim of the investigators was to develop a psychological self-help tool using modern technological means in line with the recent Femtech (female technology) developments. The hypothesis was that an online meditation tool would be more accessible and easier to integrate into a busy schedule than standard programs that require weekly attendance.

In 2017, the investigators created collaboration between experts in reproductive medicine, experts in mindfulness and a start-up that offers an online platform for meditation programs. The investigators developed an online program of 15 meditations specifically dedicated to infertile women. These meditations help women explore certain themes such as "inner resources", "social interactions", "letting go of beliefs" etc. This program has been available online since December 2017 and has been used by several thousand women.

The hypothesis behind the study is that "mindfulness-based interventions" can be delivered successfully through modern technologies with a significant impact on psychological outcomes and well-being. Femtech self-help online tools are used by thousands of women on a daily basis but studies are lacking on their efficacy.

The aim is to conduct a randomized controlled trial on the effect of a mindfulness-based intervention using the online meditation program versus standard care without intervention on psychological outcomes in infertile women undergoing ART treatments.

Women in the intervention group will receive an introduction to the concept and philosophy of mindfulness meditation through an online video and an exercise book. They will receive an access code to the application and will have access to short guided meditations both general and specific to their infertility. They will be instructed to follow the "découverte" (discovery) program of 8 meditations of 10 minutes and then the program "désir de parentalité" (wish to become a parent) of 15 meditations of 13 minutes each. Patients will be given access to all other meditations programs on the application and instructed to meditate with the program for at least 10-15 minutes on a daily basis using the e-tool for 1 month. The practice of meditation will be monitored by the number of connections to the applications and the time spent on the exercises. Women in the control group will have the standard care of the centre. The investigators will measure the effectiveness of the intervention on anxiety (State trait anxiety index, STAI), depression (Beck depression inventory, BDI), quality of life during ART treatments (Fertility quality of life tool, Fertiqol) and mindfulness aspects (Five facet mindfulness questionnaire, FFMQ). The investigators will also measure the impact of the intervention on biological stress measured by hair cortisol concentration. Finally, the investigators will assess the impact on the chances of pregnancy and on treatment discontinuation after 1 month.

ELIGIBILITY:
Inclusion Criteria:

Participants fulfilling all of the following inclusion criteria are eligible for the study:

* French-speaking
* Women between the ages of 18-42 years
* Scheduled for the first IVF treatment in HUG/CHUV/CPMA Lausanne
* Access to a computer/smartphone/tablet with access to internet and a valid Email address
* Informed Consent as documented by her signature on the form (Appendix Informed Consent Form)

Exclusion Criteria:

* Psychotropic medication
* Ongoing psychiatric/psychological treatment
* Known severe psychiatric co-morbidity

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety state scores | 1 month
  The primary aim of the study is to evaluate the effect of an e-tool based intervention versus standard care without intervention on anxiety state measured by the French version of state trait anxiety index in infertile women undergoing ART.
  State trait anxiety index state scores will be evaluated by completion of a questionnaire at 3 time points: baseline, at the time of the oocyte retrieval, on the day before the pregnancy test (before the results).
  A score between 31 and 36 is considered as normal score.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No